CLINICAL TRIAL: NCT05643404
Title: Effects of Isolated Left Bundle Branch Block on Maximal Functional Capacity
Brief Title: Effects of Isolated LBBB on Maximal Functional Capacity
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/061
Record Dates: First submitted 2022-11-22; First posted 2022-12-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-09

CONDITIONS: Left Bundle-Branch Block
Keywords: Functional capacity; Cardiac dyssynchrony; Myocardial deformation
MeSH Terms: conditions — Bundle-Branch Block | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Isolated LBBB: Subjects with left bundle branch block in the absence of clinically detectable heart disease
  Interventions: Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: Echocardioghaphy
- Matched controls without LBBB: Subjects without left bundle branch block and in the absence of clinically detectable heart disease
  Interventions: Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: Echocardioghaphy

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise testing — Maximal functional capacity will be evaluated using incremental and symptom-limited cardiopulmonary exercise testing (CPET) on a bicycle ergometer, beginning with a workload of 10 W and increasing gradually in a ramp protocol at 10-W increments every 1 minute. We will define maximal functional capacity as when the patient stops pedalling because of symptoms, and the respiratory exchange ratio (RER) is ≥1.1. During exercise, patients were monitored with 12-lead electrocardiogram and blood pressure measurements every 2 minutes. Gas exchange data and cardiopulmonary variables were averages of values taken every 10 seconds. Peak oxygen consumption (PeakVO2) will be defined as the highest value of oxygen consumption during the last 20 seconds of exercise.
Diagnostic Test: Echocardioghaphy — Doppler echocardiogram examinations were performed under resting conditions using 2-dimensional echocardiography. Left ventricular end-diastolic volume and left ventricular ejection fraction will be measured according to the European Society of Echocardiography

SUMMARY:
Left bundle branch block (LBBB) has been commonly associated with adverse cardiovascular (CV) events, but the effect of an isolated LBBB on maximal functional capacity is not well characterized.

The study's main objective is to evaluate the effect of LBBB on maximum functional capacity.

DETAILED DESCRIPTION:
Left bundle branch block (LBBB) has been commonly associated with adverse cardiovascular (CV) events, but the effect of an isolated LBBB on maximal functional capacity is not well characterized.

The main objective of the study is to evaluate the effect of LBBB on maximum functional capacity (objectively evaluated by the maximum oxygen consumption -VO2max- at peak exercise in a cardiopulmonary stress test -CPET-) in subjects with LBBB without known cardiovascular disease and compare these data with controls without LBBB.

This is a prospective study that will be carried out in a single centre. All patients with a diagnosis of LBBB and without evidence of structural heart disease in imaging tests will be enrolled. For each candidate with LBBB, one control without LBBB and matched for age, sex, body surface area, and daily physical activity will be selected. All included subjects will undergo a CPET and echocardiography. A sample size estimation [alpha: 0.05, power: 80%, and a clinically significant VO2max difference between groups of at least 10%] of 148 subjects (74 subjects with LBBB + 74 controls) would be necessary to test our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years old
* ECG criteria of left bundle branch block (for controls without left bundle branch block )
* Provide informed consent

Exclusion Criteria:

* Inability to perform a maximal baseline exercise test;
* Structural heart disease, valve heart disease or diastolic dysfunction estimated by two-dimensional echocardiography;
* Previous ischemic heart disease, heart failure, myocardiopathy or myocarditis
* Effort angina during cardiopulmonary exercise testing (CPET);
* Any moderate pulmonary disease;
* Anaemia
* Left ventricular ejection fraction < 55%.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 74 consecutive adults with a previous diagnosis of isolated left bundle branch block recruited from general practitioner outpatient clinics will be included.
  For each candidate with an isolated left bundle branch block, one control without a left bundle branch block and matched for age, sex, body surface area, and daily physical activity will be selected from general practitioner outpatient clinics
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption | Eligible patients will perform only one cardiopulmonary exercise testing on the first visit. Peak oxygen consumption will be evaluated during the procedure and compared to control patients.
  Peak oxygen consumption at peak exercise of a maximal symptom-limited cardiopulmonary exercise testing. Units peak oxygen consumption : mL/kg/min

SECONDARY OUTCOMES:
Left ventricular end-diastolic volume | Eligible patients will perform only one echocardiography on the first visit. Left ventricular end-diastolic volume will be assessed during the procedure and compared to control patients.
  Evaluate left ventricular end-diastolic indexed volume by echocardiography at rest. Unit: ml/m2
Left ventricular ejection fraction | Eligible patients will perform only one echocardiography on the first visit. Left ventricular ejection fraction will be assessed during the procedure and compared to control patients.
  Evaluate left ventricular ejection fraction by echocardiography at rest. Unit: %

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Palau, MD, PhD, Principal Investigator — Instituto de Investigacion Sanitaria INCLIVA
Locations (1):
- Marta Peiro, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Palau P, Dominguez E, Minguez S, Nunez G, Santas E, Garcia-Conejo C, de Amo I, Marin P, Flor C, Lopez L, Ortega L, Gabaldon-Sanchez I, de la Espriella R, Sanchis J, Nunez J. Effect of left bundle branch block on maximal functional capacity in asymptomatic individuals without structural heart disease. Rev Esp Cardiol (Engl Ed). 2025 Nov;78(11):957-966. doi: 10.1016/j.rec.2025.03.001. Epub 2025 Mar 21. English, Spanish. PMID 40122231